CLINICAL TRIAL: NCT00407017
Title: Therapeutic Variables in Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5264-T
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Cataract Surgery
MeSH Terms: interventions — Gatifloxacin; prednisolone acetate; Moxifloxacin; nepafenac; Methylprednisolone

INTERVENTIONS:
Drug: Gatifloxacin
Drug: Ketorolac LS
Drug: Pred Forte
Drug: Moxifloxacin
Drug: Nepafenac
Drug: EconoPred Plus

SUMMARY:
The purpose of this study is to compare patient outcomes in following cataract surgery in patients randomized to one of two surgical kits.

ELIGIBILITY:
Inclusion Criteria:

* Males or females scheduled to undergo cataract surgery
* Patients can be receiving monofocal IOLs only
* Likely to complete all study visits and able to provide informed consent
* Visual potential of 20/25 or better

Exclusion Criteria:

* Known contraindications to any study medication or ingredients
* Active ocular diseases or uncontrolled systemic disease
* Active ocular allergies

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center For Excellence in Eye Care
Locations (1):
- The Center for Excellence in Eye Care, Miami, Florida, United States